CLINICAL TRIAL: NCT03043326
Title: Demonstration Project on the Feasibility to Implement a Pre-Exposure Oral Prophylaxis Program in Men Who Have Sex With Other Men and Transgender Women at Risk of Acquiring HIV
Brief Title: Demonstration Project on the Feasibility to Implement PrEP in MSM and TG Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asociación Civil Impacta Salud y Educación, Peru (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: PrEP Peru
Record Dates: First submitted 2017-01-30; First posted 2017-02-06 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: HIV Prevention
Keywords: Pre-exposure Prophylaxis; MSM and transgender women
MeSH Terms: interventions — Tenofovir; Emtricitabine; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: Tenofovir Disoproxil Fumarate and Emtricitabine — This is an observational study. Pre-exposure Prophylaxis with TDF/3TC will be distributed to all participants elegible to receive PrEP.
  Other Names: TRUVADA tablets

SUMMARY:
The purpose of the study is to evaluating the acceptability, use and adherence of a pre-exposure prophylaxis (PrEP) program using the co-formulation tenofovir disoproxil fumarate 300 mg/emtricitabine 200 mg (TDF/FTC) administered daily by mouth, at four health facilities and one community-based organization providing health care services for MSM and transgender women.

This is an Observational, longitudinal, multicenter, open-label study to evaluate the acceptability, use and adherence to TDF/FTC-based PrEP in volunteer men who have sex with men and transgender women at substantial high risk of acquiring HIV, who were prescribed for PrEP , following the clinical guidelines to prevent HIV infection of the U.S. Centers for Disease Control and Prevention (2014) and the World Health Organization (2015).

Follow-up: Participants will be followed for 96 weeks (approximately two years) after the start of prophylactic treatment.

Implementation Target Population: Adults (≥18 years of age), without HIV infection diagnosis, and who were prescribed with PrEP and have a substantial risk of acquiring HIV infection according to the international guidelines for HIV prevention.

Sample Size: 1,000 participants

Implementation Sites:

1. Asociación Civil Impacta Salud y Educación, Barranco study site
2. Asociación Civil Impacta Salud y Educación, San Miguel study site
3. Asociación Civil Selva Amazónica, ACSA study site
4. Asociación Vía Libre, Vía Libre study site
5. Espacio Común, Epicentro study site

Primary Objectives:

1. Describing the acceptability and its socio-demographic and sexual behavior correlates for the use of PrEP.
2. Evaluate the persistence of the use of PrEP and its correlates with risk behaviors
3. Evaluating the adherence to the PrEP using self-reporting and pill counts

Secondary Objectives:

1. Describing the changes over time in risky sexual behavior among study participants.
2. Describing the number of participants who acquire HIV infection.
3. Evaluate the deviation of the indication of use of PrEP through self- reporting of its sale or sharing with third parties.

DETAILED DESCRIPTION:
HYPOTHESIS

1. Hypothesis 1. The use of PrEP based on daily intake of TDF/FTC is acceptable for MSM and transgender women and their acceptance correlates with knowledge of PrEP and sexual risk behavior.
2. Hypothesis 2. Adherence and duration of use of PrEP based on daily intake of TDF/FTC correlates with the level of education, socioeconomic level, knowledge of PrEP and risk behavior.

OBJECTIVES AND DESIGN OF THE STUDY

Primary Objectives:

1. Describing the acceptability and its socio-demographic and sexual behavior correlates for the use of PrEP.
2. Evaluate the persistence of the use of PrEP and its correlates with risk behaviors
3. Evaluating the adherence to the PrEP using self-reporting and pill counts

Secondary Objectives:

1. Describing the changes over time in risky sexual behavior among study participants.
2. Describing the number of participants who acquire HIV infection.
3. Evaluating the deviation of the indication of use of PrEP through self-reporting of its sale or sharing with third parties.

Study Design

This is an observational, longitudinal, multicenter, open-label study to evaluate the acceptability, use and adherence to PrEP in an MSM and transgender women population. Four nongovernmental organization health centers and one community-based organization in the cities of Lima and Iquitos will participate in this observational study. The study will enroll up to 1,000 participants (estimate of 200 participants per study site) for a period of 72 weeks (one and a half years). Each participant will be followed for up to 96 weeks (two years) after the start of PrEP. The estimated duration of the study implementation is 192 weeks (four years).

After enrollment, participants must attend an assessment visit at 4 weeks, 12 weeks and then every 12 weeks until they complete their participation in the study.

IMPLEMENTATION TARGET POPULATION

Description of the Study Population This PrEP research project will be implemented in volunteer MSM and transgender women without diagnosis of HIV infection and at risk of acquiring HIV because of their sexual behavior and prior to this observational study enrollment, be prescribed with PrEP by their primary care providers according the clinic guidelines of the U.S. CDC (2014) and the WHO ( 2015)

RESEARCH SITES

Each one of the proposed sites have the ability to meet the specific project implementation and procedures in this protocol. Their investigators have shown to comply with all national regulations, including good clinical practice and protection of human research subjects. The proposed sites have experience in providing comprehensive health care services to the target population and have additionally participated in research studies that have evaluated different strategies for HIV prevention.

Based on this profile, the sites are ideal for implementing the PrEP Demonstration Project in MSM and transgender women. The sites proposed for this project are:

1. Asociación Civil Impacta Salud y Educación, Barranco site
2. Asociación Civil Impacta Salud y Educación, San Miguel site
3. Asociación Civil Selva Amazónica, ACSA site
4. Asociación Vía Libre, Vía Libre site
5. Espacio Común (Epicentro), Epicentro site

The participation of a health facility of the Ministry of Health will be promoted given that with the information obtained in this study the cost-effectiveness of the program will be modeled to determine the feasibility of its escalation at various health centers that may be supported by public funds in the long term.

RECRUITMENT AND RETENTION

Recruitment The recruitment of volunteers for this study will be carried out through the implementation of a mass media campaign to promote the performing of HIV infection diagnostic testing. Virtual broadcast channels and social networking platforms will be used. In them messages will be placed in the form of banners or links to redirect users to the websites of the participating institutions, in which HIV testing diagnosis will be promoted during the time the study is implemented.

Retention of Participants

The retention of study participants will be governed by the following principles:

1. Warm care at each site will establish a friendly relationship between the participant and the staff in charge of care;
2. Quality care, including the established procedures, permanent and timely information to the user, as well as a short waiting time.

Since the primary objective of this project is to determine the feasibility of implementing a PrEP program in MSM and transgender women at risk of acquiring HIV, this study will not promote active retention of participants.

PRE-EXPOSURE PROPHYLAXIS TREATMENT

Formulation/Content TDF/FTC co-formulation contains a fixed TDF dose of 300 mg (equal to 245 mg of tenofovir disoproxil and 136 mg of tenofovir) and 200 mg of FTC.

Regimen and Administration Study participants will follow the prescription issued by their primary health care provider.

The PrEP medication will be provided at no cost by Gilead Sciences, Inc.

Product Dispensing After receiving a prescription signed by the primary care provider of the participant, the pharmacist of each site will be responsible for dispensing the medication to each participant at each visit. At the start of PrEP visit, the pharmacist will dispense one bottle and at the first follow-up visit (week 4) will dispense two bottles. At all subsequent visits to take place every 12 weeks, three bottles will be dispensed. All study participants will be advised that the medication should not be shared. Study participants that report the loss or theft of medications will be provided with additional medication.

Particularly for the Espacio Común site, which lacks a registered pharmacy that allows the storage and dispensing of products, medications will be dispensed at the Barranco de Asociación Civil Impacta Salud y Educación site pharmacy. In this scenario, the prescription will be issued at Espacio Común and with it, the participant will go to the pharmacy described at which the medication will be dispensed. It is important to mention that there are four blocks between the Espacio Común site and the Barranco site of Asociación Civil Impacta Salud y Educación. Given this geographical proximity, we do not consider that this is a problem for access to the study medication.

Product Accounting. The pharmacists of the Barranco and San Miguel sites of Asociación Civil Impacta Salud y Educación, Asociación Civil Selva Amazónica and Asociación Vía Libre will be responsible for maintaining complete and updated records of the accounting of products received or acquired.

All unused products will be returned to the central pharmacy of the study located at the Barranco site of Asociación Civil Impacta Salud y Educación once the project ends.

Adherence to the Study Medication. Adherence to PrEP will be made by counting the returned tablets at each of the scheduled visits and the self-reporting of medication intake using questionnaires applied by an interviewer.

ELIGIBILITY:
Inclusion Criteria:

* Be prescribed with PrEP
* Male biological sex;
* Age ≥18 years;
* Willing and able to provide written informed consent;

Exclusion Criteria:

* Signs or symptoms of acute retroviral syndrome;
* Upon enrollment, having a condition that, based on the opinion of the investigator or designee, prevents the participant from providing informed consent; makes participation in the project unsafe; complicates the interpretation of results; or somehow interferes with the achievement of project objectives

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This PrEP research project will be implemented in volunteer MSM and transgender women without diagnosis of HIV infection and at risk of acquiring HIV because of their sexual behavior and prior to this observational study enrollment, be prescribed with PrEP by their primary care providers according the clinic guidelines of the U.S. CDC (2014) and the WHO ( 2015)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-01-23 (Actual); Primary Completion 2020-01-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability, use and adherence of a pre-exposure prophylaxis (PrEP) program using the co-formulation tenofovir disoproxil fumarate 300 mg/emtricitabine 200 mg (TDF/FTC) administered daily by mouth, | through study completion, an average of 4 years
  At all study visits, a Computer Assisted Self Interview will be performed and get information about acceptability, self reported adherence. Pharmacist at each site will get information counting pills to measure adherence.

SECONDARY OUTCOMES:
Evaluating the deviation of the indication of use of PrEP through self-reporting of its sale or sharing with third parties. | through study completion, an average of 4 years
  Information will be captured at each visit, using CASI
Describing the changes over time in risky sexual behavior among study participants. | through study completion, an average of 4 years
  At all study visits, the Computer Assisted Self Interview will be performed and information regarding the risk behavior will be obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Gonzales, M.D., M.A.S., Study Chair — Asociación Civil Impacta Salud y Educación, Peru
Locations (5):
- Peru (5):
  - Asociacion Civil Selva amazonica, Iquitos, Maynas
  - Asociacion Via Libre, Lima
  - Asociacion Civil Impacta Salud y Educacion- Barranco CRS, Lima
  - Epicentro, Lima
  - Asociación Civil Impacta Salud y Educación-San Miguel CRS, Lima

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Grant RM, Lama JR, Anderson PL, McMahan V, Liu AY, Vargas L, Goicochea P, Casapia M, Guanira-Carranza JV, Ramirez-Cardich ME, Montoya-Herrera O, Fernandez T, Veloso VG, Buchbinder SP, Chariyalertsak S, Schechter M, Bekker LG, Mayer KH, Kallas EG, Amico KR, Mulligan K, Bushman LR, Hance RJ, Ganoza C, Defechereux P, Postle B, Wang F, McConnell JJ, Zheng JH, Lee J, Rooney JF, Jaffe HS, Martinez AI, Burns DN, Glidden DV; iPrEx Study Team. Preexposure chemoprophylaxis for HIV prevention in men who have sex with men. N Engl J Med. 2010 Dec 30;363(27):2587-99. doi: 10.1056/NEJMoa1011205. Epub 2010 Nov 23. PMID 21091279
- [Result] Anderson PL, Glidden DV, Liu A, Buchbinder S, Lama JR, Guanira JV, McMahan V, Bushman LR, Casapia M, Montoya-Herrera O, Veloso VG, Mayer KH, Chariyalertsak S, Schechter M, Bekker LG, Kallas EG, Grant RM; iPrEx Study Team. Emtricitabine-tenofovir concentrations and pre-exposure prophylaxis efficacy in men who have sex with men. Sci Transl Med. 2012 Sep 12;4(151):151ra125. doi: 10.1126/scitranslmed.3004006. PMID 22972843